CLINICAL TRIAL: NCT05243368
Title: Evaluation of Personalized Nutritional Intervention Together With the Application of MSC-derived Exosomes on the Regenerative Capacity and Wound Healing of Cutaneous Ulcers in Diabetics
Brief Title: Evaluation of Personalized Nutritional Intervention on Wound Healing of Cutaneous Ulcers in Diabetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PI21/01935
Record Dates: First submitted 2022-01-20; First posted 2022-02-17 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Foot, Diabetic
Keywords: Dietary Supplementations; Wound Healing; Diabetes Mellitus; Malnutrition
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Intervention (NI) (Experimental): In addition to the usual treatment, will receive dietary advice and a nutritional supplement, according to the results of their evaluation in the Endocrinology Service
  Interventions: Dietary Supplement: Personalized Nutritional Intervention
- Control (C) (No Intervention): Who will continue with their usual treatments in the Diabetic Foot Unit and they will receive dietary advice

INTERVENTIONS:
Dietary Supplement: Personalized Nutritional Intervention — Those with malnutrition criteria will also receive a nutritional supplement (e.g. fortimel cubitan, advanced or extra, Nutricia) or another of similar composition, in case of intolerance to the first option. The aim will be to provide at least 50% of the recommended intakes for the main nutrients related to wound healing.
  Arms: Nutritional Intervention (NI)

SUMMARY:
The ageing population and the increase in diabetes raise the prevalence of chronic skin ulcers (CCU). In diabetics, precursor cell mobilization decreases. In wounds, the inflammation is prolonged and oxidative stress increases. This is an unfavorable microenvironment for healing. A major risk factor in the development of CCU is nutritional deficiency. Healing needs energy and nutrients for regeneration. In diabetics the malnutrition can be more than 60%. However, although the provision of certain nutrients can improve the healing capacity, it is not a common clinical practice to nutritionally evaluate diabetic with CCU. Exosomes are extracellular vesicles that reflect the physiological state of the cells producing them. Stem cell derivatives exosomes are rich in factors, that can provide a favorable microenvironment for tissue regeneration.

The aim of this project is to develop a therapeutic process to accelerate the healing of diabetic CCU, based on the correction of nutritional deficiencies, to improve the regenerative capacity, together with the application of exosomes from mesenchymal stem-cell (MSC) in the wound, creating a microenvironment that favors tissue regeneration. For this, a pilot clinical trial with diabetic patients with CCU is proposed, to evaluate the effect of personalized nutritional supplementation on healing and regenerative capacity.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the informed consent
* Age between 50 and 80 years
* Diagnosis of Diabetes Mellitus for more than 1 year
* Documented diagnosis of peripheral artery disease
* HbA1c < 9%
* Category 5 in the Rutherford-Becker classification

Exclusion Criteria:

* Poor cognitive function, dementia or psychiatric conditions
* Osteomyelitis, gangrene, malignancy or immunocompromised disease
* Thromboangiitis obliterans or Buerger's disease
* Clinical evidence of invasive infection in the target limb requiring IV antibiotherapy
* Presence of neuropathic ulcers only
* Human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV) positive.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ulcer evaluation | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in size ulcer assessed by picture, including ruler to measure their size

SECONDARY OUTCOMES:
Composite measure of markers of nutritional status | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in nutritional status assessed from blood samples
Composite measure of haemogram | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in haemogram assessed from blood samples
Hemoglobin A1c (HbA1c) Test for Diabetes | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in HbA1c (%) assessed from blood samples
Measure of markers of nutritional status, include to thyrotropin | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in thyrotropin (mlU/L) assessed from blood samples
Ultrasensitive C-reactive Protein (CRP) test | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in CRP (mg/L) assessed from blood samples
Quantification of circulating endothelial progenitor cells (EPC) | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in total CD34+ or CD133+ cells expressing vascular endothelial growth factor receptor 2 (VEGFR2) analyzed by flow cytometry
Concentration of stromal cell-derived factor 1 (SDF-1) and vascular endothelial growth factor A (VEGFA) | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in concentration of SDF-1 and VEGFA factors in serum by ELISA

OTHER OUTCOMES:
Nutritional Risk | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in nutritional risk assessed by Malnutrition Universal Screening Tool (MUST)
Diagnosis of malnutrition | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in diagnosis of malnutrition assessed by Global Leadership Initiative on malnutrition (GLIM criteria)
Sarcopenia | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in sarcopenia assessed by SARC-F
Handgrip Strength | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in handgrip strength assessed by dynamometry
Body weight and height | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Body weight and height will be combined to report body mass index (BMI) in kg/m^2. Change from baseline in BMI
Tricipital skinfold | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in tricipital skinfold using a skinfold caliper
Arm circumference | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in arm circumference in centimeters (cm)
Waist and hip circumferences | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  waist and hip circumferences (cm) will be combined to report Waist and Hip Ratio (WHR). Change from baseline in WHR
Body Fat | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in body fat assessed by multifrequency bioimpedaciometry and bioelectrical impedance vector analysis
Muscle Mass | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in muscle mass assessed by multifrequency bioimpedaciometry and bioelectrical impedance vector analysis
Hydration status | Baseline, 30 days after treatment initiation, 60 days after treatment initiation and 90 days after treatment initiation
  Change from baseline in hydration status assessed by multifrequency bioimpedaciometry and bioelectrical impedance vector analysis

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Casado-Díaz, PhD, Principal Investigator — Maimonides Biomedical Research Institute of Cordoba; Alfonso Calañas, PhD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía de Córdoba, Córdoba, Andalusia, Spain

REFERENCES:
- [Background] Armstrong DG, Hanft JR, Driver VR, Smith AP, Lazaro-Martinez JL, Reyzelman AM, Furst GJ, Vayser DJ, Cervantes HL, Snyder RJ, Moore MF, May PE, Nelson JL, Baggs GE, Voss AC; Diabetic Foot Nutrition Study Group. Effect of oral nutritional supplementation on wound healing in diabetic foot ulcers: a prospective randomized controlled trial. Diabet Med. 2014 Sep;31(9):1069-77. doi: 10.1111/dme.12509. Epub 2014 Jun 19. PMID 24867069
- [Background] Basiri R, Spicer MT, Levenson CW, Ormsbee MJ, Ledermann T, Arjmandi BH. Nutritional Supplementation Concurrent with Nutrition Education Accelerates the Wound Healing Process in Patients with Diabetic Foot Ulcers. Biomedicines. 2020 Aug 3;8(8):263. doi: 10.3390/biomedicines8080263. PMID 32756299
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats A, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee; GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. Clin Nutr. 2019 Feb;38(1):1-9. doi: 10.1016/j.clnu.2018.08.002. Epub 2018 Sep 3. PMID 30181091
- [Background] Haughey L, Barbul A. Nutrition and Lower Extremity Ulcers: Causality and/or Treatment. Int J Low Extrem Wounds. 2017 Dec;16(4):238-243. doi: 10.1177/1534734617737639. Epub 2017 Nov 16. PMID 29145757
- [Background] Kurian SJ, Miraj SS, Benson R, Munisamy M, Saravu K, Rodrigues GS, Rao M. Vitamin D Supplementation in Diabetic Foot Ulcers: A Current Perspective. Curr Diabetes Rev. 2021;17(4):512-521. doi: 10.2174/1573399816999201012195735. PMID 33045979
- [Background] Malmstrom TK, Morley JE. SARC-F: a simple questionnaire to rapidly diagnose sarcopenia. J Am Med Dir Assoc. 2013 Aug;14(8):531-2. doi: 10.1016/j.jamda.2013.05.018. Epub 2013 Jun 25. No abstract available. PMID 23810110
- [Background] Zhang SS, Tang ZY, Fang P, Qian HJ, Xu L, Ning G. Nutritional status deteriorates as the severity of diabetic foot ulcers increases and independently associates with prognosis. Exp Ther Med. 2013 Jan;5(1):215-222. doi: 10.3892/etm.2012.780. Epub 2012 Oct 30. PMID 23251271